CLINICAL TRIAL: NCT06431022
Title: The Feasibility, Acceptability, and Initial Effectiveness of Web-administered Skills Training in Affective and Interpersonal Regulation (webSTAIR) for Posttraumatic Stress Disorder (PTSD) for Patients on Behavioral Health Waitlists
Brief Title: Web-administered STAIR for Patients on Behavioral Health Waitlists
Acronym: webSTAIR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H-44467
Record Dates: First submitted 2024-05-22; First posted 2024-05-28 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Post Traumatic Stress Disorder
Keywords: Digital mental health intervention (DMHI); Community health worker (CHW); Web-administered Skills Training in Affective and Interpersonal Regulation (webSTAIR); Stepped care
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-directed webSTAIR (Experimental): Participants on the Research, and Education Center (RESTORE) waitlist randomized to this arm will receive the self-managed web-administered Skills Training in Affective and Interpersonal Regulation (webSTAIR).
  Interventions: Behavioral: webSTAIR
- webSTAIR with coaching from a Community Health Worker (CHW) (Active Comparator): Participants on the RESTORE waitlist randomized to this arm will receive the web-administered Skills Training in Affective and Interpersonal Regulation (webSTAIR) with coaching support from a CHW.
  Interventions: Behavioral: webSTAIR; Behavioral: CHW coaching

INTERVENTIONS:
Behavioral: webSTAIR — WebSTAIR is a self-paced, brief skills-focused treatment for PTSD that focused on improving one's ability to manage emotions and relationships.
Behavioral: CHW coaching — CHWs will provide webSTAIR coaching, which includes motivational, problem solving, and cognitive-behavioral strategies to enhance skills practice and engagement.
  Arms: webSTAIR with coaching from a Community Health Worker (CHW)

SUMMARY:
Posttraumatic stress disorder (PTSD) is a significant public health challenge with population prevalence rates in the US between 6.1 to 9.2%. There are large racial and socioeconomic inequities in access to PTSD treatment, as up to half (30-50%) of patients in safety net clinical settings meet criteria for PTSD, yet only 13% receive any behavioral health treatment. Workforce shortages are one major barrier to accessing care. Additional barriers to care can include heightened mental health stigma and mistrust of health services.

Digital mental health interventions (DMHIs) may be suitable within the continuum of care for PTSD in hospital settings, given their potential for rapid-access, scalability, and the high acceptability of DMHI among individuals with high stigma and social needs. Among the available DMHIs for PTSD, the investigators have selected web-administered Skills Training in Affective and Interpersonal Regulation (webSTAIR), based on emerging scientific evidence and a close collaboration with Boston Medical Center (BMC) users (patients and providers) in a previous pilot study in primary care.

The aim of this randomized study is to implement webSTAIR at BMC in the Recovery from Stress and Trauma through Outpatient Care, Research, and Education (RESTORE) Center's subspecialty clinic.

ELIGIBILITY:
Inclusion Criteria:

* Client on the RESTORE Center waitlist at Boston Medical Center
* Over 18 years of age
* Able to receive therapy in English or Spanish (per participant report)
* Exposure to trauma (as indicated by the Life Events Checklist for the DSM-5 [LEC-5])
* Probable PTSD (as indicated by the PTSD Checklist for the DSM-5 [PCL-5] based on PCL score of 33+).
* Reasonable to access to technology (e.g., phone, computer, internet access).

Exclusion Criteria:

* Patient declines to be in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2024-11-15 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Feasibility based on recruitment rate | 3 months
  The recruitment rate will be calculated by dividing the number of participants by the total number of eligible participants.
Feasibility based on assessment completion rate | 3 months, 6 months
  The proportion of assessments completed will be calculated by dividing the number of assessments completed by the total number of participants.
Feasibility based on attendance rate | 3 months
  The attendance rate will be calculated by dividing the number of webSTAIR sessions attended by the potential number of webSTAIR sessions for each participant.
Client satisfaction | 3 months, 6 months
  Client satisfaction/acceptability will be measured by the Client Satisfaction Questionnaire (CSQ-8) which is an 8 item instrument with each item having 4 potential responses form 1 to 4. Scores are summed across items once. Items 2, 4, 5, and 8 are reverse scored. Total scores range from 8 to 32, with the higher number indicating greater satisfaction.

SECONDARY OUTCOMES:
PTSD Checklist for DSM-5 (PCL-5) | baseline, 3 months, 6 months
  The PCL-5 is a 20-item self-report checklist of PTSD symptoms based on the DSM-5 criteria1. It measures the degree to which respondents have been bothered by each symptom over the past month or week. To score the PCL-5, a cut-off raw score of 38 is used for a provisional diagnosis of PTSD. Additionally, the DSM-5 diagnostic rule requires at least one symptom from cluster B (questions 1-5), one from cluster C (questions 6-7), two from cluster D (questions 8-14), and two from cluster E (questions 15-20).
Trauma Symptoms of Discrimination (TSDS) | baseline, 3 months, 6 months
  The Trauma Symptoms of Discrimination Scale (TSDS) is a 21 item self-report measure designed to assess the traumatizing impact of discrimination broadly by measuring anxiety-related symptoms of trauma due to discriminatory experiences. Participants report the frequency of their experience of discriminatory distress regarding trauma on a 4-point scale ranging from 0 (Never) to 3 (Often). Scores can range from 0 to 63 and higher scores are associated with more trauma symptoms of discrimination.
Work and Social Functioning (WSAS) | baseline, 3 months, 6 months
  The WSAS is scored using a 9-point Likert-type scale ranging from 0 (no impairment) to 8 (severe impairment). Potential scores range from 0 to 40 with higher scores indicating higher levels of impairment in the assessed areas of a respondent's life.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Valentine, PhD, Principal Investigator — Boston Medical Center, Psychiatry Department
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No